CLINICAL TRIAL: NCT01566942
Title: FOLFIRI or mFOLFOX6 as Adjuvant Chemotherapy Regiment After Neo-adjuvant Chemotherapy With FOLFIRI in Patients With Advanced Colorectal Cancer: a Randomized, Multicenter Clinical Trial
Brief Title: FOLFIRI or mFOLFOX6 in Adjuvant Chemotherapy in Advanced Colorectal Cancer
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Sun Yat-sen University (Other)
Collaborators: First Affiliated Hospital, Sun Yat-Sen University (Other)
Responsible Party: Principal Investigator, Yulong He, GI Surgery, the First Affiliated Hospital, Sun Yat-sen University, Sun Yat-sen University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2011-170
Record Dates: First submitted 2012-03-26; First posted 2012-03-30 (Estimated); Last update posted 2012-03-30 (Estimated); Status verified 2012-03

CONDITIONS: Colorectal Cancer
Keywords: FOLFIRI; FOLFOX; adjuvant chemotherapy; advanced colorectal cancer
MeSH Terms: conditions — Colorectal Neoplasms | interventions — Oxaliplatin; Irinotecan

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- FOLFOX (Active Comparator): In this group, the patients will receive the adjuvant chemotherapy with mFOLFOX6.
  Interventions: Drug: Oxaliplatin
- FOLFIRI (Experimental): in this arm, patients will receive adjuvant chemotherapy with FOLFIRI regimen for about 8 cycles
  Interventions: Drug: Irinotecan

INTERVENTIONS:
Drug: Oxaliplatin — In this arm, patients will receive the adjuvant chemotherapy with mFOLFOX6 regimen for 8 cycles. Oxaliplatin 85mg/m2, day1, every 2 weeks; Leucovorin 200mg/m2,day1,every 2 weeks;5-FU 400mg/m2,iv, day1, 5-FU 3.0g/m2, bolus for 46h,every 2 weeks
  Arms: FOLFOX
Drug: Irinotecan — In this arm, patients will receive the adjuvant chemotherapy with FOLFIRI regimen for 8 cycles. Irinotecan 180mg/m2, day1, every 2 weeks; Leucovorin 200mg/m2,day1,every 2 weeks;5-FU 400mg/m2,iv, day1, 5-FU 3.0g/m2, bolus for 46h,every 2 weeks
  Arms: FOLFIRI

SUMMARY:
the aim of this study is to observe the effect of irinotecan-based regimen in patients with advanced colorectal cancer.

ELIGIBILITY:
Inclusion Criteria:

* histologically confirmed adenocarcinoma in colorectal cancer
* clinical stage Ⅲ or Ⅳa(with potential radical resective metastatic lesions),≥ 12 lymph nodes examined
* no cancer cells were found in ascites
* Eastern Cooperative Oncology Group(ECOG) performance status of 0-2
* male or female, between 18 and 75 years old
* adequate hematologic, hepatic and renal functions
* without severe heart disease in the last 6 months before enrolled. If with hypertension or coronary artery disease, it can be controlled
* not enrolled into others clinical trial during this study
* all patients should sign the informed consent

Exclusion Criteria:

* can not be tolerated operation
* receiving others therapy(including Traditional Chinese herbs)for this disease, can not obey the investigator during the study
* can not be tolerated the adverse effect of drugs in these regimens
* major surgery within 4 weeks prior to study treatment start, or lack of complete recovery from major surgery
* metastatic disease more than one organ
* pregnant or lactating women

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2012-06; Primary Completion 2014-05 (Estimated); Study Completion 2017-06 (Estimated)

PRIMARY OUTCOMES:
disease-free survival（DFS） | 3-year disease-free survival rate
  The investigator will follow up all the enrolled patients. The difference of 3-year-DFS between two groups will be compared.

SECONDARY OUTCOMES:
overall survival(OS) | 5-year survival
  The 5-year survival rate will be the secondary end point. The investigator will follow up the patients and campare the difference of 5-year-OS between the two groups.

CONTACTS AND LOCATIONS:
Overall Officials: YULONG HE, PhD, Study Chair — First Affiliated Hospital, Sun Yat-Sen University
Locations (1):
- the first affiliated hospital of Sun Yat-sen University, Guangzhou, Guangdong, China